CLINICAL TRIAL: NCT03289364
Title: A Phase 2 Study to Assess the Safety and Efficacy of Scalp Cooling Using PenguinTM Cold Caps for the Prevention or Reduction of Chemotherapy-induced Alopecia in Stage I-III Breast Cancer
Brief Title: Penguin Cold Caps in the Prevention of Hair Loss in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Providence Health & Services (Other)
Collaborators: Medical Specialties of California (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017000277
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Alopecia; Hair Loss; Scalp Cooling; Penguin Cold Caps
MeSH Terms: conditions — Breast Neoplasms; Alopecia

STUDY DESIGN:
Intervention Model Description: Patients will use the Penguin Cold Caps during prior to, during, and after chemotherapy administration. Cold-cap therapy will commence at least 50 minutes prior to infusion, and will continue for 4 hours following completion of chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penguin Cold Caps (Experimental): Penguin Cold-cap therapy will commence at least 50 minutes prior to chemotherapy infusion, and will continue for 4 hours following completion of chemotherapy.
  Interventions: Device: Penguin Cold Caps

INTERVENTIONS:
Device: Penguin Cold Caps — Patients will wear Penguin Cold Cap scalp cooling device prior to each chemotherapy administration, during administration, and for four hours following administration.

SUMMARY:
The goal of this study is to estimate the efficacy of Penguin cold caps in preventing or reducing hair loss in patients receiving (neo)adjuvant chemotherapy (one of four common regimens) for early stage breast cancer.

DETAILED DESCRIPTION:
This will be a phase II prospective, open label, non-randomized study conducted to determine the safety and efficacy of Penguin TM cold cap system in preventing or reducing chemotherapy-induced alopecia in patients with early stage breast cancer undergoing chemotherapy.

Eligible subjects will be enrolled to one of 4 study arms (Table 5) determined by type of chemotherapy. Subjects will have early stage breast cancer of any receptor subtype, for which standard of care includes chemotherapy. Eligible subjects will be enrolled at Providence Portland Medical Center (PPMC) and Providence St. Vincent Medical Center (PSVMC).

The PenguinTM cold cap therapy will be administered to all enrolled subjects according to the dosing schedule specified by the study arms. PenguinTM cold caps is a portable scalp cooling system which uses gel-filled cold caps that are cooled on dry ice and exchanged every 30 minutes in order to maintain optimum temperature. Its unique crylon gel formula is specifically created to maintain cold temperatures for much longer periods of time than other conventional cooling gels and foams. No scalp preparation is required before use.

ELIGIBILITY:
Inclusion Criteria:

* At least ≥ 18 years of age
* Diagnosis of stage I-III breast cancer for whom neoadjuvant or adjuvant cytotoxic chemotherapy (ACT/HP, TCH/P, TC, or T/H) is planned.
* Willing and able to provide informed consent.
* Availability of caretaker(s) to accompany participant and facilitate cold-cap placement/exchanges using the recommended technique.
* Women of childbearing potential must use acceptable measures to avoid becoming pregnant during study period and for 30 days after last dose of chemotherapy.

Exclusion Criteria:

* Pre-existing alopecia (Dean's scale ≥ 1)
* Another malignancy that required active treatment with systemic chemotherapy within 2 years of study recruitment.
* Prior radiotherapy treatment involving head.
* Pre-existing chronic severe headaches or migraines.
* Skin conditions that in the opinion of PI would be at risk of worsening with study.
* Cold sensitivity or cold agglutinin disease
* Cryoglobulinemia
* Cryofibrogenemia
* History of current evidence of any condition, therapy or abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, such that trial participation is not in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Deans Alopecia Scale | 30 days post chemotherapy treatment
  Number of patients who score from 0-2 on Deans Alopecia Scale

SECONDARY OUTCOMES:
Was it Worth it Questionnaire | 30 days post chemotherapy treatment
  Number of patients reporting positive or beneficial effects of Cold Cap therapy on the Was it Worth it Questionnaire.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 | 30 days post chemotherapy treatment
  Number of patients reporting positive or beneficial effects of Cold Cap therapy on the EORTC QLQ-C30
Body Image Scale Questionnaire | 30 days post chemotherapy treatment
  These outcomes will be reported as the proportion of patients (and confidence intervals) reporting the study cold-cap therapy as positive and beneficial on the Body Image Scale Questionnaire
Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 30 days post chemotherapy treatment
  The proportion of patients (and confidence intervals) with grade 1 or 2 alopecia according to CTCAE rating scale

CONTACTS AND LOCATIONS:
Overall Officials: David Page, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Cancer Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No